CLINICAL TRIAL: NCT00059761
Title: Phase I Study of Irinotecan and Cisplatin in Combination With Twice Daily Thoracic Radiotherapy (45 Gy) or Once Daily Thoracic Radiotherapy (70 Gy) for Patients With Limited Stage Small Cell Lung Cancer
Brief Title: Chemotherapy Combined With Radiation Therapy in Treating Patients With Limited-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0241; CDR0000269348
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; Irinotecan; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Sequence A: Level 1 (Experimental): Irinotecan 40 mg/m2, cisplatin 60 mg/m2, concurrent radiation therapy (RT) at 1.5 Gy BID
  Interventions: Drug: cisplatin; Drug: irinotecan hydrochloride; Radiation: radiation therapy
- Sequence B: Level 1 (Experimental): Irinotecan 40 mg/m2, cisplatin 60 mg/m2, concurrent RT at 2 Gy once daily
  Interventions: Drug: cisplatin; Drug: irinotecan hydrochloride; Radiation: radiation therapy
- Sequence A: Level 2 (Experimental): Irinotecan 50 mg/m2, cisplatin 60 mg/m2, concurrent radiation therapy (RT) at 1.5 Gy BID
  Interventions: Drug: cisplatin; Drug: irinotecan hydrochloride; Radiation: radiation therapy
- Sequence B: Level 2 (Experimental): Irinotecan 50 mg/m2, cisplatin 60 mg/m2, concurrent RT at 2 Gy once daily
  Interventions: Drug: cisplatin; Drug: irinotecan hydrochloride; Radiation: radiation therapy
- Sequence A: Level 3 (Experimental): Irinotecan 60 mg/m2, cisplatin 60 mg/m2, concurrent radiation therapy (RT) at 1.5 Gy BID
  Interventions: Drug: cisplatin; Drug: irinotecan hydrochloride; Radiation: radiation therapy
- Sequence B: Level 3 (Experimental): Irinotecan 60 mg/m2, cisplatin 60 mg/m2, concurrent RT at 2 Gy once daily
  Interventions: Drug: cisplatin; Drug: irinotecan hydrochloride; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin
Drug: irinotecan hydrochloride
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effect on the body when combining irinotecan and cisplatin with radiation therapy in treating patients who have limited-stage small cell lung cancer that could not be completely removed during surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of irinotecan administered with cisplatin and thoracic radiotherapy (given at two different schedules) in patients with limited stage small cell lung cancer.
* Determine the qualitative and quantitative toxicity and non-dose-limiting toxicity of these regimens in these patients.
* Determine the reversibility of all toxic effects associated with these regimens in these patients.

OUTLINE: This is a non-randomized, dose-escalation study of irinotecan. Patients are assigned to 1 of 2 radiotherapy (RT) treatment groups.

* Radiotherapy:

  * Group I: Patients undergo thoracic RT twice daily, 5 days a week, for 3 weeks.
  * Group II: Patients undergo thoracic RT once daily, 5 days a week, for 7 weeks.
* Concurrent chemotherapy: Patients receive irinotecan IV over 60-90 minutes on days 1 and 8 and cisplatin IV over 1 hour on day 1. Treatment repeats every 3 weeks for 1 course for group I and 2 courses for group II.
* Post RT chemotherapy: Patients receive irinotecan and cisplatin as above for 3 courses for group I and 2 courses, beginning after RT is complete, for group II.

Sequential cohorts of 6 patients per group receive escalating doses of irinotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 3 months for 1 year and then 6 months for 4 years.

PROJECTED ACCRUAL: A total of 12-36 patients (6-18 per group) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell lung cancer by one of two methods:

  * Fine needle aspiration biopsy
  * Two positive sputa
* Must have limited disease as defined by all of the following:

  * Stage I-IIIB
  * Confined to 1 hemithorax
  * No T4 tumor based on malignant pleural or pericardial effusion

    * Patients with pleural effusion too small to tap under CT guidance and not evident on chest x-ray are allowed
  * No N3 disease based on contralateral hilar or contralateral supraclavicular involvement
* Measurable or evaluable disease

  * Tumor must be able to be encompassed by specified radiotherapy fields without unacceptable risk of serious pulmonary compromise
* No complete tumor resection
* No pericardial effusion (regardless of cytology)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 120,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* No known Gilbert's disease

Renal

* Creatinine no greater than 1.5 mg/dL

Cardiovascular

* No myocardial infarction within the past 6 months
* No symptomatic heart disease

Pulmonary

* Forced expiratory volume (FEV)_1 at least 1.0 L/sec
* No uncontrolled bronchospasms
* No uncompensated chronic obstructive pulmonary disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No pre-existing peripheral neuropathy grade 2 or greater
* No other malignancy within the past 2 years except curatively treated basal or squamous cell skin cancer or carcinoma in situ of the bladder or cervix
* No other concurrent serious medical illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic therapy

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy
* No concurrent intensity-modulated radiotherapy

Surgery

* See Disease Characteristics

Other

* At least 7 days since prior enzyme-inducing anti-convulsant drugs (EIACDs) (e.g., phenytoin, carbamazepine, or phenobarbital) if used on a regular basis for more than 2 weeks

  * Less than 2 weeks of regular use of EIACDs does not require a 7-day wash-out period
* At least 14 days since prior Hypericum perforatum (St. John's wort)
* No concurrent EIACDs
* No concurrent amifostine during chemoradiotherapy
* Concurrent gabapentin or other non-EIACDs allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2003-03; Primary Completion 2009-03 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of irinotecan in combination with cisplatin and thoracic radiotherapy (45 Gy BID or 70 Gy daily) by toxicity assessment (Common Toxicity Criteria version 3.0) during acute and late toxicity | From the start of treatment until 90 days

SECONDARY OUTCOMES:
Rate of non-dose limiting toxicity | From start of treatment to the end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Corey J. Langer, MD, Study Chair — Fox Chase Cancer Center; Maria Werner-Wasik, MD, Study Chair — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (49):
- United States (49):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Saint Rose Hospital, Hayward, California
  - Valley Memorial Hospital, Livermore, California
  - Highland General Hospital at St. George's University School of Medicine, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Summit Medical Center, Oakland, California
  - J.C. Robinson, M.D. Regional Cancer Center, San Pablo, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Michael & Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Wendt Regional Cancer Center at Finley Hospital, Dubuque, Iowa
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Monmouth Medical Center, Long Branch, New Jersey
  - Fox Chase Virtua Health Cancer Program - Marlton, Mount Holly, New Jersey
  - AtlantiCare Regional Medical Center, Pomona, New Jersey
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Mercy Cancer Institute at Mercy Hospital, Pittsburgh, Pennsylvania
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - Greenville Hospital System Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Sarah Cannon Cancer Center at Parkridge Medical Center, Chattanooga, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin

REFERENCES:
- [Result] Langer CJ, Swann S, Werner-Wasik M, et al.: Phase I study of irinotecan (Ir) and cisplatin (DDP) in combination with thoracic radiotherapy (RT), either twice daily (45 Gy) or once daily (70 Gy), in patients with limited (Ltd) small cell lung carcinoma (SCLC): early analysis of RTOG 0241. [Abstract] J Clin Oncol 24 (Suppl 18): A-7058, 378s, 2006.
- [Result] Langer C, Swann S, Werner-Wasik M, et al.: Phase I study of combination irinotecan and cisplatin and either twice daily thoracic radiation (45Gy) or once daily thoracic radiotherapy (70Gy) in patients with limited small cell lung carcinoma (SCLC): early toxicity analysis of RTOG 0241. [Abstract] Lung Cancer 49 (Suppl 2): A-P-777, S323, 2005.